CLINICAL TRIAL: NCT07281716
Title: A Phase 1b/2 Study of Combination Immunotherapy for the Treatment of Chemotherapy-refractory Metastatic Microsatellite Stable (MSS) Colorectal Cancer (CRC)
Brief Title: Combination Immunotherapy for the Treatment of Chemotherapy-refractory Metastatic MSS CRC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dan Feng (Other)
Collaborators: Coherus Oncology, Inc. (Industry); Cantargia AB (Industry)
Responsible Party: Sponsor-Investigator, Dan Feng, Assistant Professor in Medicine, Hematology and Medical Oncology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-25-00756; PRMC-25-046 IIT (Other: PRMC)
Record Dates: First submitted 2025-11-25; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Microsatellite Stable Colorectal Carcinoma
Keywords: Colorectal Cancer(CRC); Chemotherapy-refractory colorectal cancer; Microsatellite stable colorectal cancer (MSS CRC); Metastatic colorectal cancer; Chemotherapy-resistant CRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: 3+3 run-in subjects, first 3 subjects will be enrolled and the first constitutes the DLT window. If there are 2 or more subjects experiencing a DLT, the trial will be halted and the treatment plan discussed with the Tisch Cancer Institute DSMC. If 0 or 1 subject experience a DLT, 3 more subjects will be enrolled. If 2+ subjects experience a DLT the trial will be halted and the treatment plan discussed with the DSMC. If at most 1 out of 6 subjects experiences a DLT, Phase 2 of the trial will open. The 6 subjects from the Phase 1b portion will be evaluable as part of the Phase 2 cohort of 21 subjects and will follow a two-stage minimax design, with 12 subjects in Stage 1 and 9 subjects in Stage 2. A safety stopping rule for futility will be applied and expect that 10% of participants could be expected to drop out either in the phase 1b or phase 2 and will be replaced. Therefore, the total number of subjects that could be enrolled in order to obtain 21 evaluable subjects will be 24
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nadunolimab and Toripalimab (Experimental): Participants will receive the investigational combination of nadunolimab and toripalimab. Treatment will continue for up to 1 year or until disease progression, whichever occurs first.
  Interventions: Drug: Nadunolimab; Drug: Toripalimab

INTERVENTIONS:
Drug: Nadunolimab — 5 mg/kg intravenously (IV) every 3 weeks (Q3W)
Drug: Toripalimab — 240 mg IV every 3 weeks (Q3W)

SUMMARY:
Phase 1b/2 open-label study evaluates the safety, tolerability, and efficacy of combination immunotherapy with nadunolimab (anti-IL-1RAP) and toripalimab (anti-PD-1) in patients with chemotherapy-refractory metastatic microsatellite stable (MSS) colorectal cancer. Phase 1b will assess dose-limiting toxicity (DLT), while Phase 2 will evaluate objective response rate (ORR), including progression-free survival (PFS), overall survival (OS), disease control rate (DCR), and duration of response (DOR). Exploratory analyses will investigate immunomodulatory effects through tumor and peripheral blood studies, and treatment will continue every 3 weeks for up to 1 year or until disease progression.

DETAILED DESCRIPTION:
This is a Phase 1b/2, open-label study evaluating the safety, tolerability, and efficacy of nadunolimab (anti-IL-1RAP) in combination with toripalimab (anti-PD-1) in adults with chemotherapy-refractory metastatic microsatellite stable (MSS) colorectal cancer. The Phase 1b portion serves as a safety run-in with up to 6 subjects to assess the safety of a single dose of the combination therapy. Following this, Phase 2 will enroll up to 21 subjects, with the first 6 from Phase 1b included in the Phase 2 analysis to assess the primary efficacy endpoint. Eligible participants must have biopsy-confirmed MSS colorectal cancer (non-MSI-high or pMMR), whose disease has progressed during or following 5-FU, oxaliplatin and/or irinotecan-based chemotherapy with or without a biological agent. Subjects must have have measurable disease and tumor accessible for core needle biopsy. Participants will receive nadunolimab 5 mg/kg and toripalimab 240 mg intravenously every three weeks, continuing for up to one year or until disease progression. Primary objectives: For Phase 1/b, to determine the safety and tolerability of combination immunotherapy in subjects with chemotherapy-refractory metastatic non-MSI-high/pMMR CRC. For Phase 2, to determine the efficacy of combination immunotherapy in subjects with chemotherapy-refractory metastatic non-MSI-high/pMMR CRC as measured by the objective response rate (ORR) achieved. Subjects will undergo core needle biopsies, blood collection, and repeat imaging throughout the study. This study is conducted at Mount Sinai Hospital under IRB and PRMC oversight. The results will provide important information on the safety and potential efficacy of combining nadunolimab and toripalimab in a population with limited treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathologically confirmed diagnosis of non-MSI-H/pMMR CRC.
* Patients must have progressed (clinically or radiographically) on or after standard chemotherapy, including fluoropyrimidines, oxaliplatin, and irinotecan, or are intolerant to standard chemotherapy. Patients may have received, if eligible, anti-VEGF or anti-EGFR antibodies in combination with chemotherapy.
* Patients must have at least 1 measurable target lesion at baseline ≥ 10mm in the longest diameter.
* Patient must be willing and able to provide blood samples (6 heparinized, and two streck tubes, roughly 70 - 80 mL) at the time points indicated in the Study Calendar.
* Patients must have at least 1 lesion suitable for core needle biopsies.
* Patients must be willing and able to have core needle biopsies, if clinically feasible (Goal 3-6 biopsies, final number to be determined by the interventionalist performing the procedure as safe), of tumor prior to initiation of study drug. Should patients undergo pre-treatment or on-treatment biopsy procedure and inadequate number of biopsies are obtained, they may proceed with initiation/continuation of treatment at the discretion of the investigator and treating physician.
* Age ≥ 18 years.
* ECOG Performance Status 0-1 (Karnofsky ≥60%, see https://ecog-acrin.org/resources/ecog-performance-status/). o Patients with performance status >1 carrying long-term disability (such as cerebral palsy) where the disability is not acute nor progressive, and unlikely to significantly affect their response to therapy may be enrolled at the investigator's discretion
* Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 4 months following completion of therapy. Should a study participant become pregnant or suspect pregnancy while participating in this study, the study participant should inform the treating physician immediately. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: o Has not undergone a hysterectomy or bilateral oophorectomy; or o Has not been naturally postmenopausal for at least 12 consecutive months
* Ability to understand and the willingness to sign a written informed consent. • Adequate organ and marrow function

Exclusion Criteria:

* Patients who have had chemotherapy within 14 days from start of therapy.
* Palliative radiotherapy is permitted at anytime, if deemed in the best interest of the patient.
* Patients may not be receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring antibiotics (exception is a brief (≤10days) course of antibiotics to be completed before initiation of treatment), symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who have undergone major surgery within 4 weeks prior to the first dose of treatment.
* Patients who are pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Patients who discontinued prior immune checkpoint inhibitors due to immune-related adverse events are not eligible for enrollment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Patients on chronic steroids (more than 4 weeks at stable dose) equivalent to ≤ 10mg prednisone will not be excluded.
* Has active autoimmune disease that has required systemic treatment in the past 1 year (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is acceptable.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
* HIV positive with detectable viral load, or anyone not on stable anti-viral (HAART) regimen, or with <200 CD4+ T cells/microliter in the peripheral blood. HIV testing is mandatory for patients with no known history of HIV. For such patients HIV testing will be considered SOC.
* Has known active Hepatitis B (e.g., HBV detected by PCR or active Hepatitis C (e.g., HCV RNA [qualitative] is detected). Patients with hepatitis B (HepBsAg+) who have controlled infection (serum hepatitis B virus DNA PCR that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA. Patients must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study drug.
* History of allogeneic hematopoietic cell transplantation or solid organ transplantation.
* Receipt of a live vaccine within 28 days of planned start of study medication.
* Receipt of etanercept or other TNF-α inhibitors within 28 days of planned start of the study medication.
* Documented allergic or hypersensitivity response to any protein therapeutics (e.g., recombinant proteins, vaccines, intravenous immune globulins, monoclonal antibodies, receptor traps).
* Principal investigator believes that for one or multiple reasons the patient will be unable to comply with all study visits, or if they believe the trial is not clinically in the best interest of the patient.
* History of irAE in response to prior immunotherapy that has not improved to a Grade 0 or 1; this does not include chronic conditions such as endocrinopathies which can be treated with hormone replacement therapy.
* History of interstitial lung disease (e.g., idiopathic pulmonary fibrosis, organizing pneumonia) or active, noninfectious pneumonitis attributed to prior use of cancer immunotherapy that required immune-suppressive doses of glucocorticoids to assist with management. A history of radiation pneumonitis in the radiation field is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities (DLTs) | The first cycle (day1 - day21) constitutes the DLT window.
  For the Phase 1b portion, Dose-Limiting Toxicities (DLTs) will be assessed based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. Adverse events are graded on a scale from 1 (mild) to 5 (death related to AE). Permanent discontinuation of study treatment will occur for any severe (Grade 3) drug-related adverse event that recurs or for any life-threatening (Grade 4) event.
Objective Response Rate (ORR) | Treatment initiation through 12 months, or until documented disease progression or initiation of new anti-cancer therapy, whichever occurs first
  For the phase 2 portion, ORR will be assessed based on the definition, as the combined percent of the subjects experiencing a partial response (PR) or a complete response (CR) at anytime within the first year from the initiation of therapy, or until the documented progression of disease or start of a new anti-cancer therapy. Radiographic response will be determined by the RECIST v1.1

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | From first dose through disease progression, death, or up to 12 months, whichever occurs first.
  Progression-free survival (PFS) is defined as the time in days from the first administration of nadunolimab until documented progression of disease on imaging or death.
Overall survival (OS) | From first administration of nadunolimab until documented death from any cause, or up to 12 months, whichever occurs first.
  Overall survival (OS) is defined as the time in days from the first administration of nadunolimab until documented death from any cause.
Disease control rate (DCR) | From first administration of nadunolimab until best objective response, or up to 12 months, whichever occurs first.
  Disease control rate (DCR) is defined as the percent of the subjects experiencing a best objective response of PR, CR or stable disease (SD).
Duration of response (DOR) | up to 12 months
  Duration of response (DOR) is defined as the time from which a subject achieves either a PR or a CR until subsequent progression of disease is documented radiographically or clinically.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Feng, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The completed dataset is the sole property of the Sponsor-Investigator's institution and should not be exported to third parties, except for authorized representatives of appropriate Health/Regulatory Authorities, without permission from the Sponsor-investigator and their institution.

REFERENCES:
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Prager GW, Taieb J, Fakih M, Ciardiello F, Van Cutsem E, Elez E, Cruz FM, Wyrwicz L, Stroyakovskiy D, Papai Z, Poureau PG, Liposits G, Cremolini C, Bondarenko I, Modest DP, Benhadji KA, Amellal N, Leger C, Vidot L, Tabernero J; SUNLIGHT Investigators. Trifluridine-Tipiracil and Bevacizumab in Refractory Metastatic Colorectal Cancer. N Engl J Med. 2023 May 4;388(18):1657-1667. doi: 10.1056/NEJMoa2214963. PMID 37133585
- [Background] Benson AB, Venook AP, Al-Hawary MM, Arain MA, Chen YJ, Ciombor KK, Cohen S, Cooper HS, Deming D, Farkas L, Garrido-Laguna I, Grem JL, Gunn A, Hecht JR, Hoffe S, Hubbard J, Hunt S, Johung KL, Kirilcuk N, Krishnamurthi S, Messersmith WA, Meyerhardt J, Miller ED, Mulcahy MF, Nurkin S, Overman MJ, Parikh A, Patel H, Pedersen K, Saltz L, Schneider C, Shibata D, Skibber JM, Sofocleous CT, Stoffel EM, Stotsky-Himelfarb E, Willett CG, Gregory KM, Gurski LA. Colon Cancer, Version 2.2021, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2021 Mar 2;19(3):329-359. doi: 10.6004/jnccn.2021.0012. PMID 33724754
- [Background] Pages F, Mlecnik B, Marliot F, Bindea G, Ou FS, Bifulco C, Lugli A, Zlobec I, Rau TT, Berger MD, Nagtegaal ID, Vink-Borger E, Hartmann A, Geppert C, Kolwelter J, Merkel S, Grutzmann R, Van den Eynde M, Jouret-Mourin A, Kartheuser A, Leonard D, Remue C, Wang JY, Bavi P, Roehrl MHA, Ohashi PS, Nguyen LT, Han S, MacGregor HL, Hafezi-Bakhtiari S, Wouters BG, Masucci GV, Andersson EK, Zavadova E, Vocka M, Spacek J, Petruzelka L, Konopasek B, Dundr P, Skalova H, Nemejcova K, Botti G, Tatangelo F, Delrio P, Ciliberto G, Maio M, Laghi L, Grizzi F, Fredriksen T, Buttard B, Angelova M, Vasaturo A, Maby P, Church SE, Angell HK, Lafontaine L, Bruni D, El Sissy C, Haicheur N, Kirilovsky A, Berger A, Lagorce C, Meyers JP, Paustian C, Feng Z, Ballesteros-Merino C, Dijkstra J, van de Water C, van Lent-van Vliet S, Knijn N, Musina AM, Scripcariu DV, Popivanova B, Xu M, Fujita T, Hazama S, Suzuki N, Nagano H, Okuno K, Torigoe T, Sato N, Furuhata T, Takemasa I, Itoh K, Patel PS, Vora HH, Shah B, Patel JB, Rajvik KN, Pandya SJ, Shukla SN, Wang Y, Zhang G, Kawakami Y, Marincola FM, Ascierto PA, Sargent DJ, Fox BA, Galon J. International validation of the consensus Immunoscore for the classification of colon cancer: a prognostic and accuracy study. Lancet. 2018 May 26;391(10135):2128-2139. doi: 10.1016/S0140-6736(18)30789-X. Epub 2018 May 10. PMID 29754777
- [Background] Diakos CI, Charles KA, McMillan DC, Clarke SJ. Cancer-related inflammation and treatment effectiveness. Lancet Oncol. 2014 Oct;15(11):e493-503. doi: 10.1016/S1470-2045(14)70263-3. PMID 25281468
- [Background] Mantovani A, Allavena P, Sica A, Balkwill F. Cancer-related inflammation. Nature. 2008 Jul 24;454(7203):436-44. doi: 10.1038/nature07205. PMID 18650914
- [Background] Binnewies M, Roberts EW, Kersten K, Chan V, Fearon DF, Merad M, Coussens LM, Gabrilovich DI, Ostrand-Rosenberg S, Hedrick CC, Vonderheide RH, Pittet MJ, Jain RK, Zou W, Howcroft TK, Woodhouse EC, Weinberg RA, Krummel MF. Understanding the tumor immune microenvironment (TIME) for effective therapy. Nat Med. 2018 May;24(5):541-550. doi: 10.1038/s41591-018-0014-x. Epub 2018 Apr 23. PMID 29686425
- [Background] Sondalle SB, Baserga SJ. Ribosomes Need Straight A's to Sleep. Cell. 2017 May 4;169(4):565-567. doi: 10.1016/j.cell.2017.04.019. PMID 28475888
- [Background] Kenny PJ, Zhou H, Kim M, Skariah G, Khetani RS, Drnevich J, Arcila ML, Kosik KS, Ceman S. MOV10 and FMRP regulate AGO2 association with microRNA recognition elements. Cell Rep. 2014 Dec 11;9(5):1729-1741. doi: 10.1016/j.celrep.2014.10.054. Epub 2014 Nov 20. PMID 25464849
- [Background] Salmon H, Idoyaga J, Rahman A, Leboeuf M, Remark R, Jordan S, Casanova-Acebes M, Khudoynazarova M, Agudo J, Tung N, Chakarov S, Rivera C, Hogstad B, Bosenberg M, Hashimoto D, Gnjatic S, Bhardwaj N, Palucka AK, Brown BD, Brody J, Ginhoux F, Merad M. Expansion and Activation of CD103(+) Dendritic Cell Progenitors at the Tumor Site Enhances Tumor Responses to Therapeutic PD-L1 and BRAF Inhibition. Immunity. 2016 Apr 19;44(4):924-38. doi: 10.1016/j.immuni.2016.03.012. PMID 27096321
- [Background] Garris CS, Arlauckas SP, Kohler RH, Trefny MP, Garren S, Piot C, Engblom C, Pfirschke C, Siwicki M, Gungabeesoon J, Freeman GJ, Warren SE, Ong S, Browning E, Twitty CG, Pierce RH, Le MH, Algazi AP, Daud AI, Pai SI, Zippelius A, Weissleder R, Pittet MJ. Successful Anti-PD-1 Cancer Immunotherapy Requires T Cell-Dendritic Cell Crosstalk Involving the Cytokines IFN-gamma and IL-12. Immunity. 2018 Dec 18;49(6):1148-1161.e7. doi: 10.1016/j.immuni.2018.09.024. Epub 2018 Dec 11. PMID 30552023
- [Background] Coussens LM, Zitvogel L, Palucka AK. Neutralizing tumor-promoting chronic inflammation: a magic bullet? Science. 2013 Jan 18;339(6117):286-91. doi: 10.1126/science.1232227. PMID 23329041
- [Background] Lv Y, Cao D, Guo F, Qian Y, Wang C, Wang D. Abdominal wall reconstruction using a combination of free tensor fasciae lata and anterolateral thigh myocutaneous flap: a prospective study in 16 patients. Am J Surg. 2015 Aug;210(2):365-73. doi: 10.1016/j.amjsurg.2014.11.008. Epub 2015 Mar 5. PMID 25824825
- [Background] LaMarche NM, Hegde S, Park MD, Maier BB, Troncoso L, Le Berichel J, Hamon P, Belabed M, Mattiuz R, Hennequin C, Chin T, Reid AM, Reyes-Torres I, Nemeth E, Zhang R, Olson OC, Doroshow DB, Rohs NC, Gomez JE, Veluswamy R, Hall N, Venturini N, Ginhoux F, Liu Z, Buckup M, Figueiredo I, Roudko V, Miyake K, Karasuyama H, Gonzalez-Kozlova E, Gnjatic S, Passegue E, Kim-Schulze S, Brown BD, Hirsch FR, Kim BS, Marron TU, Merad M. An IL-4 signalling axis in bone marrow drives pro-tumorigenic myelopoiesis. Nature. 2024 Jan;625(7993):166-174. doi: 10.1038/s41586-023-06797-9. Epub 2023 Dec 6. PMID 38057662
- [Background] Rizvi NA, Hellmann MD, Snyder A, Kvistborg P, Makarov V, Havel JJ, Lee W, Yuan J, Wong P, Ho TS, Miller ML, Rekhtman N, Moreira AL, Ibrahim F, Bruggeman C, Gasmi B, Zappasodi R, Maeda Y, Sander C, Garon EB, Merghoub T, Wolchok JD, Schumacher TN, Chan TA. Cancer immunology. Mutational landscape determines sensitivity to PD-1 blockade in non-small cell lung cancer. Science. 2015 Apr 3;348(6230):124-8. doi: 10.1126/science.aaa1348. Epub 2015 Mar 12. PMID 25765070
- [Background] Snyder A, Makarov V, Merghoub T, Yuan J, Zaretsky JM, Desrichard A, Walsh LA, Postow MA, Wong P, Ho TS, Hollmann TJ, Bruggeman C, Kannan K, Li Y, Elipenahli C, Liu C, Harbison CT, Wang L, Ribas A, Wolchok JD, Chan TA. Genetic basis for clinical response to CTLA-4 blockade in melanoma. N Engl J Med. 2014 Dec 4;371(23):2189-2199. doi: 10.1056/NEJMoa1406498. Epub 2014 Nov 19. PMID 25409260
- [Background] Coughlan JJ, Wafer M, Fitzgerald G, Nawaz A, O'Brien C, Liston R. QTc prolongation in acute medical admissions: an often overlooked and potentially serious finding. Postgrad Med J. 2018 Feb;94(1108):123-124. doi: 10.1136/postgradmedj-2017-135208. Epub 2017 Sep 28. No abstract available. PMID 28972097
- [Background] Tesio M, Trinquand A, Ballerini P, Hypolite G, Lhermitte L, Petit A, Ifrah N, Baruchel A, Dombret H, Macintyre E, Asnafi V. Age-related clinical and biological features of PTEN abnormalities in T-cell acute lymphoblastic leukaemia. Leukemia. 2017 Dec;31(12):2594-2600. doi: 10.1038/leu.2017.157. Epub 2017 May 25. PMID 28539671
- [Background] Larsen CH. The fragile environments of inexpensive CD4+ T-cell enumeration in the least developed countries: strategies for accessible support. Cytometry B Clin Cytom. 2008;74 Suppl 1:S107-16. doi: 10.1002/cyto.b.20386. PMID 18228565
- [Background] Anthony B. El-Khoueiry et al. Results from a phase 1a/1b study of botensilimab (BOT), a novel innate/adaptive immune activator, plus balstilimab (BAL; anti-PD-1 antibody) in metastatic heavily pretreated microsatellite stable colorectal cancer (MSS CRC).. J Clin Oncol 41, LBA8-LBA8(2023).